CLINICAL TRIAL: NCT03928288
Title: Novel, Non-Hormonal Therapy for the Treatment of Chronic Pain Due to Endometriosis in Adolescent and Adult Women
Brief Title: Cabergoline for the Treatment of Chronic Pain Due to Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Thomas Jefferson University (Other); Stanford University (Other); Children's Hospital Colorado (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Amy DiVasta, MD, Associate Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00031528
Record Dates: First submitted 2019-04-04; First posted 2019-04-26 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Cabergoline 0.5 mg PO twice weekly for 6 months
  Interventions: Drug: Cabergoline 0.5 MG
- Placebo (Placebo Comparator): Placebo capsule PO twice weekly for 6 months
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: Cabergoline 0.5 MG — Medication
  Other Names: Dostinex
  Arms: Intervention
Drug: Placebo - Cap — Placebo capsule
  Arms: Placebo

SUMMARY:
Endometriosis is dependent on angiogenesis (the sprouting of new blood vessels) for its growth and maintenance, but the side effects of currently approved angiogenesis inhibitors make these agents inappropriate for use in reproductive-age patients. This obstacle will be overcome by performing a randomized, double blind clinical trial aimed at repurposing an existing drug, cabergoline, as a safe, alternative angiogenesis inhibitor for adolescents and young women with endometriosis. This trial proposes a novel, non-hormonal, non-surgical therapeutic approach aimed at alleviating the pain and suffering associated with this common chronic disease that currently has limited treatment options.

DETAILED DESCRIPTION:
Endometriosis is a gynecologic condition in which tissue similar to the inside lining of the uterus (the endometrium) grows in locations in the body outside of the uterus. This abnormal growth can cause severe pain, often coinciding with a woman's menstrual period. Endometriosis affects about 10% of all women of reproductive age in the US, and leads to an estimated $22 billion/year in health care costs in the US alone. Endometriosis is a chronic disease that can progress over time, leading to infertility, debilitating pelvic pain, and resulting poor quality of life. Disease management involves not only prompt initiation of therapy, but also the maintenance of therapy for a prolonged length of time. As no cure currently exists, the disease typically progresses until menopause. Current medical management typically consists of hormonal medications and surgery, but these therapies are limited by lack of successful relief of symptoms, cost, or side effects. Many patients have endometriosis pain that is refractory to all available treatments. Safe, well-tolerated, long-duration additions to currently available treatments are sorely needed to ameliorate the chronic course of this disease.

Angiogenesis refers to the generation of new blood vessels from existing vessels. It is required for the growth of new living tissue and has been implicated in the initiation, maintenance, and spread of endometriosis. The investigators hypothesize that medications that inhibit the process of angiogenesis can be used to treat endometriosis. The angiogenesis inhibitor medications that are currently available cause severe side effects such as birth defects that prevent them from being safely used for treating endometriosis in young, otherwise healthy women. In contrast, there is an alternative medication, cabergoline, which has been extensively used in clinical practice for treatment of other endocrine conditions suffered by reproductive-aged women. While cabergoline appears to inhibit angiogenesis, it acts on this process indirectly such that it has very few side effects, making it appropriate for use in young women with endometriosis.

The investigators will conduct a clinical drug trial to determine whether cabergoline is an effective addition to standard hormonal therapy for decreasing persistent pelvic pain suffered by adolescents and young women with surgically-proven endometriosis. Patients who are interested in participating in our study will be randomized (decided by a flip of a coin) to either receive cabergoline, the investigational medication, or a placebo pill (a sugar pill). It is believed that after 6 months, patients who take cabergoline twice a week will demonstrate decreased pain scores and improved quality of life/ability to perform daily activities as compared to patients who take a placebo pill (sugar pill) twice weekly. During the research study, the investigators will study how pain symptoms, menstrual bleeding, levels of inflammation, risk for future cardiac disease, and measures of pain sensitivity change over time by using well-established, validated tools and techniques that the research team has utilized successfully in previous work.

ELIGIBILITY:
Inclusion Criteria:

* Female with surgically-confirmed endometriosis
* Age 15 years to 40 years
* Current use ≥ 2 months duration of hormonal therapy such as combined oral contraceptives, norethindrone acetate, or levonorgestrel intrauterine device
* Current pelvic pain (score ≥ 3 on Visual Analog Scale, where 0 represents absence of pain and 10 indicates unbearable pain) present for ≥ 14 days/month over the 2 months prior to study enrollment
* Willingness to comply with visit schedule and protocol

Exclusion Criteria:

* Pre-menarche or post-menopause
* Contraindications to cabergoline (e.g., cardiac valve disorder; pulmonary, pericardial, retroperitoneal fibrotic disorder; hypersensitivity to ergot derivatives; uncontrolled hypertension)
* Significant mental or chronic systemic illness that might confound pain assessment or the ability to complete the study
* Pregnant, breastfeeding, or planning to become pregnant in the next 6 months
* Impaired liver function (ALT > 2x normal) or liver disease
* Breast cancer, current or previous
* Thromboembolic disease, current or previous
* Use of other drugs that affect dopamine (e.g., phenothiazines, metoclopramide, butyrophenones)

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 129 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Change in pain assessed by the Brief Pain Inventory Interference Scale (BPI) over 6 months | every 6 weeks for 6 months
  BPI: A 7-item self-report measure. The items in this scale can be grouped into those that assess physical functioning (general activity; walking ability; normal work, including both work outside the home and housework), those that assess emotional functioning (mood; relations with people; enjoyment of life), and a single item that assesses the extent to which pain interferes with sleep. Either the item asking about the "worst pain" or the arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference. The BPI is anchored between a scale of zero (no pain/interference) to ten (maximum pain/interference). The magnitude of treatment-associated change in BPI Interference Scale scores in open-label and randomized clinical trials ranges from 1 to 3 points, depending on the specific pain conditions and treatments studied.
Change in pain severity measured by Visual Analog Scale (VAS) over 6 months | every 6 weeks for 6 months
  VAS: A measurement of pain intensity, assessed by a 0 to 10 numerical rating scale, to rate maximum and average pain intensity over the preceding 7 days. Higher scores indicate more severe pain intensity.
Change in pain measured by Biberoglu and Behrman patient ratings scale (B&B pain scale) over 6 months | every 6 weeks for 6 months
  Biberoglu and Behrman patient ratings scale (B&B pain scale): Survey that assesses dyspareunia, dysmenorrhea, and noncyclic pelvic pain. Each is graded on a scale from 0 to 3 (or 4), with higher numbers indicating more severe symptoms.

SECONDARY OUTCOMES:
Change in measurements of serum biomarkers of angiogenesis and inflammation over 6 months | every 3 months for 6 months
  Measurement of serum concentrations of high sensitivity C-reactive protein, interleukins 1B and 8, tumor necrosis factor alpha, and vascular endothelial growth factor
Change in cardiovascular dysfunction measured by pulse wave velocity over 6 months | baseline and 6 months
  Peripheral wave velocity is an ultrasound measurement of the rate at which pressure waves move down a blood vessel. It is collected by using two pressure catheters placed a known distance from one another, the "Pulse Wave Distance".
Change in measures of central hypersensitization measured by quantitative sensory testing at 6 months | every 3 months for 6 months
  Quantitative sensory testing (QST) is a single, standardized protocolized test that involves measurement of 3 pain threshold tests (cutaneous dynamic brush allodynia, muscular pain threshold, temporal summation test) that will be measured at the abdomen
Incidence of vaginal bleeding over 6 months | completed daily for 6 months
  Measurement of the incidence of vaginal bleeding using phone-based survey to document the presence/absence of vaginal bleeding

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Standford University, Palo Alto, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania